CLINICAL TRIAL: NCT04745026
Title: An Exploratory, Phase 2, Randomized, Double-blind, Placebo-controlled Trial to Investigate the Safety and Efficacy of Cannabidiol Oral Solution (GWP42003-P; CBD-OS) in Children and Adolescents With Autism Spectrum Disorder
Brief Title: Trial to Investigate the Safety and Efficacy of Cannabidiol Oral Solution (GWP42003-P; CBD-OS) in Children and Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWND19189; 2020-002819-21 (EudraCT Number)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Cannabidiol oral solution; CBD-OS; GWP42003-P; Children; Adolescents
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GWP42003-P 10 mg/kg/day (Experimental): Participants will be stratified based on their age (6 to 11 years old, 12 to 17 years old), use of antipsychotics (on versus off), and region (North America versus Rest of the World) and will be randomized to receive 5 milligrams per kilogram per day (mg/kg/day) GWP42003-P for 1 week and then 10 mg/kg/day GWP42003-P for 11 weeks.
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Participants will be stratified based on their age (6 to 11 years old, 12 to 17 years old), use of antipsychotics (on versus off), and region (North America versus Rest of the World) and will be randomized to receive matching placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P — GWP42003-P oral solution (100 milligrams per milliliter [mg/mL] cannabidiol [CBD] in sesame oil with anhydrous ethanol, ethanol [10% v/v] sweetener [sucralose], and strawberry flavoring), administered twice a day (morning and evening)
  Other Names: Epidiolex®; cannabidiol; CBD-OS
  Arms: GWP42003-P 10 mg/kg/day
Drug: Placebo — Oral placebo to match GWP42003-P oral solution containing sesame oil with anhydrous ethanol, sweetener (sucralose), strawberry flavoring, and beta carotene, administered twice a day (morning and evening)
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the efficacy of GWP42003-P, compared with placebo, in reducing symptom severity in children with Autism Spectrum Disorder (ASD).

ELIGIBILITY:
Inclusion Criteria:

* Participant weight is at least 12 kilograms (kg).
* Participants (if possessing adequate understanding, in the investigator's opinion) and their parent(s)/legal representative are willing and able to give informed assent and consent for participation in the trial.
* Participant and their caregiver are willing and able (in the investigator's opinion) to comply with all trial requirements.
* Participant has a diagnosis of Autism Spectrum Disorder (ASD) as per Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for ASD, confirmed by Autism Diagnostic Observational Schedule (ADOS-2) criteria (conducted within 2 years at the trial site or at screening by a qualified assessor). Note: During special circumstances (e.g., COVID-19 pandemic) where the ADOS-2 cannot be performed due to site restrictions (e.g., mandatory use of face masks) and an ADOS- 2 conducted within 2 years at the trial site by a qualified assessor is not available, eligibility can be confirmed using: 1) an ADOS-2 performed within 2 years by a qualified assessor (external to the site); 2) if 1) is not available, eligibility may be confirmed using the Autism Diagnostic Interview, Revised (ADI-R) at screening.
* Clinical Global Impressions - Improvement Scale (CGI-S) ≥ 4 (moderately ill) at screening and randomization.
* Intelligence quotient (IQ) ≥ 70 at screening, or measured within 1 year of screening, using Wechsler Abbreviated Scale of Intelligence Scale Second Edition (WASI-II).
* All medications or interventions (including psychosocial interventions, dietary supplements, probiotics, speech therapy, etc.) for ASD related symptoms must have been stable for 4 weeks prior to screening and randomization, and the patient/caregiver should be willing to maintain a stable regimen throughout the trial.
* Participants must have the ability to swallow the investigational medicinal product (IMP), provided as a liquid solution.
* Participant and/or parent(s)/legal representative is willing to allow the responsible authorities to be notified of participation in the trial, if mandated by local law.
* Participant and/or parent(s)/legal representative is/are willing to allow the participant's primary care practitioner (if they have one) and consultant (if they have one) to be notified of participation in the trial if the primary care practitioner/consultant is different from the investigator.

Exclusion Criteria:

* Current diagnosis of bipolar disorder, psychosis, schizophrenia, schizoaffective disorder, or major depression (participants with depression in remission may be included)
* Has a diagnosis other than ASD that dominates the clinical presentation (e.g., Attention Deficit Hyperactivity Disorder [ADHD])
* Has a progressive neurological condition
* Seizures in the past 24 weeks
* Changes in anticonvulsive therapy within the last 12 weeks
* Currently taking more than 2 anti-epileptic drugs (AEDs)
* Taking sirolimus, everolimus, temsirolimus, or tacrolimus
* Taking clobazam
* Taking omeprazole, lansoprazole, tolbutamide, or warfarin
* Taking repaglinide, pioglitazone, rosiglitazone, montelukast, bupropion, or efavirenz
* Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®, or Epidiolex®) within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP, such as sesame oil.
* Participant has moderately impaired hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) or total bilirubin (TBL) > 2 × ULN. This criterion can only be confirmed once the laboratory results are available; participants enrolled into the trial who are later found to meet this criterion must be screen-failed.
* Participant is male and fertile (i.e., after puberty unless permanently sterile by bilateral orchidectomy) unless willing to ensure that they use male contraception (condom) or remain sexually abstinent during the trial and for 12 weeks thereafter.
* Participant is female and of childbearing potential (i.e., following menarche and until becoming postmenopausal for ≥ 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that they use a highly effective method of birth control (e.g., hormonal contraception, intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence) during the trial and for 12 weeks thereafter.
* Female participant who is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the trial or within 12 weeks thereafter.
* Participant has received an IMP within the 12 weeks prior to the screening visit.
* Participant had brain surgery or traumatic brain injury within 1 year of screening.
* Participant has any other significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.
* Any abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if they took part in the trial
* Any history of suicidal behavior (lifelong) or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 4 weeks or at screening or randomization
* Participant has donated blood during the past 12 weeks and is unwilling to abstain from donation of blood during the trial.
* Participant has any known or suspected history of alcohol or substance abuse or positive drugs of abuse test at screening (not justified by a known concurrent medication).
* Participant has previously been randomized into this trial.
* Participant has plans to travel outside their country of residence during the trial, unless the participant has confirmation that the IMP is permitted in the destination country/state

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (12):
  - Southwest Autism Research and Resource Center (SARRRC), Phoenix, Arizona
  - UCSD School of Medicine, La Jolla, California
  - UCLA Neuropsychiatric Institute, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - APG Research, LLC, Orlando, Florida
  - University of Louisville, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital (Lurie Center for Autism), Lexington, Massachusetts
  - Richmond Behavioral Associates, Staten Island, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Seattle Children's Research Institute, Seattle, Washington
- Australia (2):
  - Monash Medical Centre, Clayton
  - Queensland Children's Hospital, South Brisbane
- Canada (2):
  - The Kids Clinic, Ajax, Ontario
  - Center for Pediatric Excellence, Ottawa, Ontario
- Germany (2):
  - Klinik fur Psychiatrie, Psychotherapie und Psychosomatik im Kindes und Jugendalter, Freiburg im Breisgau
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim
- Spain (3):
  - Instituto Global de Atencion Integral del Neurodesarrollo (IGAIN), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell
- United Kingdom (2):
  - University of Glasgow Institute of Health and Wellbeing, Glasgow
  - Institute of Psychiatry, King's College London, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 191 patients were screened for this study. Of those 191 patients, 103 patients met all inclusion criteria and no exclusion criteria were enrolled in the study and randomized to treatment at 24 centers in the United States, Canada, Spain, United Kingdom, and Australia.
Pre-assignment Details: Eligible participants were randomized 7 to 14 days after the screening visit (Visit 1), once all required assessments were completed and laboratory results were reviewed. If required, screening assessments were permitted to be split over 2 visits; however, both visits were conducted within 7- to 14-day window prior to randomization (Visit 2).
Groups:
- GWP42003-P: Patients who were randomized to 5 mg/kg/day GWP42003-P for 1 week and then 10 mg/kg/day GWP42003-P for 11 weeks. At the end of treatment, participants tapered off the medication over a period of 1 week.
- Placebo: Patients who were randomized to placebo for 12 weeks.
Period: Overall Study
Arm/Group | GWP42003-P | Placebo
Started | 49 | 54
Completed | 36 | 41
Not Completed | 13 | 13
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P | Placebo | Total
Number analyzed (Participants) | 49 | 54 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 54 | 103
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (3.02) | 10.8 (3.01) | 10.9 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 36 | 47 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 2 | 3
  Black or African American | 5 | 2 | 7
  White | 32 | 42 | 74
  Multiple | 5 | 2 | 7
  Unknown | 2 | 1 | 3
  Not Reported | 1 | 2 | 3
  Other | 2 | 1 | 3
WASI-II Intelligent Quotient Score [Mean (Standard Deviation); unit: score on a scale] — Population: The WASI-II raw score is converted into T-scores and then summed to derive the composite score, which ranges from 70 (worst outcome) to 160 (best outcome). Composite score performance categories are: Profoundly high=150-160, Superior= 130-160, Very high=120-129, Bright normal=110-119, Average=90-109, Low average=80-89, and Borderline=70-79.
  score on a scale | 99.42 (18.03) | 100.89 (17.16) | 100.19 (17.49)
Aberrant Behavior Checklist Irritability [Mean (Standard Deviation); unit: score on a scale] — On the Aberrant Behavior Checklist (ABC), the irritability score is based on a 15-item subscale where each item is rated on a 4-point scale, ranging from 0 (not a problem) to 3 (severe problem). The total score ranges from 0 to 45, with higher scores indicating worst clinical outcome and lower scores indicating better clinical outcome. Population: Aberrant Behavior Checklist Irritability was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 54 | 102
    (all) | 23.2 (7.36) | 22.5 (8.74) | 22.8 (8.09)
Aberrant Behavior Checklist Social Withdrawal [Mean (Standard Deviation); unit: score on a scale] — On the Aberrant Behavior Checklist (ABC), the social withdrawal score is based on a 16-item subscale where each item is rated on a 4-point scale, ranging from 0 (not a problem) to 3 (severe problem). The total score ranges from 0 to 48, with higher scores indicating worst clinical outcome and lower scores indicating better clinical outcome. Population: Aberrant Behavior Checklist Social Withdrawal was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 54 | 102
    (all) | 12.6 (8.63) | 12.7 (9.11) | 12.7 (8.85)
Aberrant Behavior Checklist Stereotypic Behavior [Mean (Standard Deviation); unit: score on a scale] — On the Aberrant Behavior Checklist (ABC), the stereotypic behavior score is based on a 7-item subscale where each item is rated on a 4-point scale, ranging from 0 (not a problem) to 3 (severe problem). The total score ranges from 0 to 21, with higher scores indicating worst clinical outcome and lower scores indicating better clinical outcome. Population: Aberrant Behavior Checklist Stereotypic Behavior was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 54 | 102
    (all) | 6.7 (5.08) | 6.7 (4.83) | 6.7 (4.92)
Aberrant Behavior Checklist Hyperactivity/Noncompliance [Mean (Standard Deviation); unit: score on a scale] — On the Aberrant Behavior Checklist (ABC), the hyperactivity/noncompliance score is based on a 16-item subscale where each item is rated on a 4-point scale, ranging from 0 (not a problem) to 3 (severe problem). The total score ranges from 0 to 48, with higher scores indicating worst clinical outcome and lower scores indicating better clinical outcome. Population: Aberrant Behavior Checklist Hyperactivity/Noncompliance was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 54 | 102
    (all) | 25.2 (12.27) | 26.9 (9.63) | 26.1 (10.93)
Aberrant Behavior Checklist Inappropriate Speech [Mean (Standard Deviation); unit: score on a scale] — On the Aberrant Behavior Checklist (ABC), the inappropriate speech score is based on a 4-item subscale where each item is rated on a 4-point scale, ranging from 0 (not a problem) to 3 (severe problem). The total score ranges from 0 to 12, with higher scores indicating worst clinical outcome and lower scores indicating better clinical outcome. Population: Aberrant Behavior Checklist Inappropriate Speech was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 54 | 102
    (all) | 5.7 (3.22) | 5.6 (3.08) | 5.6 (3.13)
Vineland Adaptive Behavior Scales Social and Communication Composite Score [Mean (Standard Deviation); unit: score on a scale] — The Vineland Social and Communication Composite Score ranges from 20 (worst clinical outcome) to 160 (best clinical outcome). Scores from 115 to 160 is above average, 86 to 114 average, 71 to 85 below average, and below 70 low. Population: Vineland Adaptive Behavior Scales Social and Communication Composite Score was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 48 | 50 | 98
    (all) | 66.6 (19.61) | 67.7 (15.18) | 67.2 (17.41)
Clinical Global Impression - Severity (CGI-S) [Mean (Standard Deviation); unit: score on a scale] — The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's experience with patients who have the same diagnosis. The clinician is asked: Considering your total clinical experience with this particular population, how ill is the patient at this time? This is rated as: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill. Higher scores indicate worse outcome. Population: Clinical Global Impression - Severity (CGI-S) was assessed in participants with available data in the Full Analysis Set.
  score on a scale
    number analyzed (Participants) | 49 | 51 | 100
    (all) | 4.76 (0.630) | 4.82 (0.684) | 4.79 (0.656)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Subscale Total Scores
Description: The caregiver-assessed ABC was designed to assess the presence and severity of various problem behaviors commonly observed in individuals diagnosed with intellectual and developmental disability. The checklist contains 5 subscales: Irritability (15 items); Social Withdrawal (16 items); Stereotypic Behavior (7 items); Hyperactivity/Noncompliance (16 items); and Inappropriate Speech (4 items). Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). The total score of all items for each subscale range from 0-45 (irritability), 0-48 (social withdrawal and hyperactivity/noncompliance), 0-21 (stereotypic behavior), and 0-12 (inappropriate speech) where higher scores indicate worse clinical outcome. The change from baseline to Week 4, Week 8, and Week 12 is reported with lower scores indicating better clinical outcome.
Time Frame: Baseline up to Week 12
Population: Aberrant behavior checklist subscale total scores were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 40 | 51
score on a scale
  ABC-Irritability, Week 4 | -6.35 (7.98) | -5.41 (7.16)
  ABC-Irritability, Week 8: number analyzed (Participants) | 36 | 43
  ABC-Irritability, Week 8 | -6.67 (8.63) | -8.05 (9.12)
  ABC-Irritability, Week 12: number analyzed (Participants) | 34 | 35
  ABC-Irritability, Week 12 | -6.97 (9.68) | -8.57 (10.10)
  ABC-Social Withdrawal, Week 4 | -2.53 (5.61) | -2.92 (5.24)
  ABC-Social Withdrawal, Week 8: number analyzed (Participants) | 36 | 43
  ABC-Social Withdrawal, Week 8 | -3.81 (6.76) | -4.74 (6.25)
  ABC-Social Withdrawal, Week 12: number analyzed (Participants) | 34 | 35
  ABC-Social Withdrawal, Week 12 | -3.74 (6.21) | -4.51 (5.95)
  ABC-Stereotypic Behavior, Week 4 | -2.10 (4.24) | -1.39 (3.24)
  ABC-Stereotypic Behavior, Week 8: number analyzed (Participants) | 36 | 43
  ABC-Stereotypic Behavior, Week 8 | -1.92 (3.99) | -1.98 (4.05)
  ABC-Stereotypic Behavior, Week 12: number analyzed (Participants) | 34 | 35
  ABC-Stereotypic Behavior, Week 12 | -1.88 (3.63) | -2.31 (4.03)
  ABC-Hyperactivity/Noncompliance, Week 4 | -5.73 (8.08) | -4.55 (8.15)
  ABC-Hyperactivity/Noncompliance, Week 8: number analyzed (Participants) | 36 | 43
  ABC-Hyperactivity/Noncompliance, Week 8 | -6.39 (9.15) | -7.42 (9.06)
  ABC-Hyperactivity/Noncompliance, Week 12: number analyzed (Participants) | 34 | 35
  ABC-Hyperactivity/Noncompliance, Week 12 | -6.74 (10.62) | -8.77 (9.94)
  ABC-Inappropriate Speech, Week 4 | -2.13 (2.88) | -0.88 (2.07)
  ABC-Inappropriate Speech, Week 8: number analyzed (Participants) | 36 | 43
  ABC-Inappropriate Speech, Week 8 | -1.58 (2.74) | -1.44 (2.73)
  ABC-Inappropriate Speech, Week 12: number analyzed (Participants) | 34 | 35
  ABC-Inappropriate Speech, Week 12 | -1.94 (2.93) | -1.51 (2.97)
Statistical Analysis 1: Comparison: GWP42003-P vs Placebo; Irritability (Week 12); Test type: Superiority; p = 0.085, Mixed models for repeated measures — Randomization factors, baseline score, visit, treatment arm, visit by treatment arm (fixed), and visit repeated within each patient (repeated); Least square mean difference = 3.37, 95% CI 2-sided [-0.48 to 7.21], Standard Error of Mean 1.931
Statistical Analysis 2: Comparison: GWP42003-P vs Placebo; Social Withdrawal Week 12); Test type: Superiority; p = 0.3107, Mixed models for repeated measures; Randomization factors, baseline score, visit, treatment arm, visit by treatment arm (fixed), and visit repeated within each patient (repeated); Least square mean difference = 1.14, 95% CI 2-sided [-1.08 to 3.36], Standard Error of Mean 1.16
Statistical Analysis 3: Comparison: GWP42003-P vs Placebo; Stereotypic Behavior (Week 12); Test type: Superiority; p = 0.9513, Mixed models for repeated measures; [statistical method as in outcome 1, analysis 2]; Least square mean difference = 0.04, 95% CI 2-sided [-1.34 to 1.42], Standard Error of Mean 0.695
Statistical Analysis 4: Comparison: GWP42003-P vs Placebo; Hyperactivity/Noncompliance (Week 12); Test type: Superiority; p = 0.305, Mixed models repeated measures; [statistical method as in outcome 1, analysis 2]; Least square mean difference = 2.01, 95% CI 2-sided [-1.86 to 5.88], Standard Error of Mean 1.943
Statistical Analysis 5: Comparison: GWP42003-P vs Placebo; Inappropriate Speech (Week 12); Test type: Superiority; p = 0.4754, Mixed models repeated measures; [statistical method as in outcome 1, analysis 2]; Least square mean difference = -0.37, 95% CI 2-sided [-1.4 to 0.66], Standard Error of Mean 0.517

2. Primary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales-3 (VABS-3) Scores
Description: The VABS-3 scales assess what a person does, rather than what he or she can do. The Vineland-3 assesses adaptive behavior in 3 domains: Communication, Daily Living Skills, and Socialization. Each domain is comprised of 3 subdomains: receptive expression and written (communication); personal, domestic and community (daily living skills); Interpersonal relationships, play and leisure and copying skills (socialization). The adaptive behavior composite score is calculated as arithmetic mean of all 3 domain scores. The total score range is 20 to 140, where low scores indicate low (worst) clinical outcome and high scores indicate high (best) clinical outcome. The change from baseline in VABS-3 is being reported with positive values indicating a positive improvement in adaptive behavior.
Time Frame: Baseline up to Week 12
Population: Vineland Adaptive Behavior Scales-3 (VABS-3) scores were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 37 | 45
score on a scale
  Week 4 | 2.97 (6.70) | 0.99 (9.29)
  Week 8: number analyzed (Participants) | 36 | 40
  Week 8 | 3.69 (10.82) | 3.54 (8.83)
  Week 12: number analyzed (Participants) | 31 | 32
  Week 12 | 4.85 (8.83) | 5.55 (10.42)
Statistical Analysis 1: Comparison: GWP42003-P vs Placebo; Week 12; Test type: Superiority; p = 0.8506, Mixed models for repeated measures; [statistical method as in outcome 1, analysis 2]; Least square mean difference = 0.45, 95% CI 2-sided [-4.26 to 5.15], Standard Error of Mean 2.36

3. Primary Outcome: Number of Patients Per Clinical Global Impression Improvement (CGI-I) Category
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. The clinician is asked: Compared to the patient's condition at admission to the project, how much has the patient changed? This is rated as: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. Higher scores indicate worse clinical outcome. The number of patients in each CGI-I category is reported.
Time Frame: Day 85
Population: Patients per CGI-I category were assessed in participants with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 34 | 38
Participants
  Minimally improved | 13 | 14
  Much improved | 12 | 11
  No change | 9 | 11
  Much worse | 0 | 1
  Very much improved | 0 | 1
  Minimally worse | 0 | 0
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: GWP42003-P vs Placebo; Responders with 'Very Much Improved' or 'Much Improved' response at week 12; Test type: Superiority; p = 0.7087, Regression, Logistic; Includes treatment arm, randomization variables and baseline score (CGI-S) covariates. Responders achieved a score of 1 or 2 at post-baseline visits; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.43 to 3.51]

4. Primary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scores
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's experience with patients who have the same diagnosis. The clinician is asked: Considering your total clinical experience with this particular population, how ill is the patient at this time? This is rated as: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill. Higher scores indicate worse outcome. The change from baseline in CGI-S scores is reported and lower mean scores indicate better outcome.
Time Frame: Baseline up to Week 12
Population: CGI-S was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 43 | 51
score on a scale
  Week 4 | -0.33 (0.61) | -0.31 (0.69)
  Week 8: number analyzed (Participants) | 40 | 42
  Week 8 | -0.50 (0.68) | -0.48 (0.92)
  Week 12: number analyzed (Participants) | 31 | 32
  Week 12 | -0.55 (0.85) | -0.63 (1.10)
Statistical Analysis 1: Comparison: GWP42003-P vs Placebo; Week 12; Test type: Superiority; p = 0.6108, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events
Description: A TEAE is one that started, or worsened in severity or seriousness, following the first dose of IMP. AEs were coded according to the Medical Dictionary for Regulatory Activities v24.0 dictionary.
Time Frame: Baseline up to Week 12
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 49 | 54
Participants
  TEAE | 27 | 24
  Non-TEAE | 25 | 32
  Treatment-related TEAE | 6 | 10
  Serious TEAE | 2 | 1
  Serious Treatment-related TEAE | 0 | 0
  TEAE leading to study intervention withdrawal | 2 | 1
  Treatment-related TEAE leading to drug withdrawal | 1 | 1
  TEAE leading to withdrawal | 2 | 2
  TEAE leading to death | 0 | 0

6. Secondary Outcome: Mean Change From Baseline in Hematology Clinical Laboratory Levels
Time Frame: Baseline up to Week 9 (end of taper/withdrawal)
Population: Hematology clinical laboratory levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 30 | 37
10^9 cells/L
  Week 9: Basophils | -0.01 (0.03) | 0 (0.03)
  Week 9: Eosinophils | -0.09 (0.311) | 0 (0.40)
  Week 9: Lymphocytes | 0.04 (0.70) | -0.20 (0.68)
  Week 9: Monocytes | -0.01 (0.15) | -0.01 (0.19)
  Week 9: Neutrophils | 0.04 (1.80) | -0.01 (1.26)
  Week 9: Platelets | -9.43 (34.50) | 8.43 (52.13)
  Week 9: Leukocytes | -0.02 (1.87) | -0.23 (1.79)

7. Secondary Outcome: Mean Percentage Change From Baseline in Hematology Clinical Laboratory Levels
Time Frame: Baseline up to Week 9 (end of taper/withdrawal)
Population: Hematology clinical laboratory levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 31 | 38
percentage change from baseline
  Week 9: Basophils/Leukocytes: number analyzed (Participants) | 30 | 37
  Week 9: Basophils/Leukocytes | -0.07 (0.45) | -0.03 (0.42)
  Week 9: Eosinophils/Leukocytes: number analyzed (Participants) | 30 | 37
  Week 9: Eosinophils/Leukocytes | -1.33 (5.37) | 0.22 (4.88)
  Week 9: Hematocrit | -0.02 (2.19) | 0.43 (2.30)
  Week 9: Lymphocytes/Leukocytes: number analyzed (Participants) | 30 | 37
  Week 9: Lymphocytes/Leukocytes | 1.05 (11.25) | -2.32 (8.26)
  Week 9: Monocytes/Leukocytes: number analyzed (Participants) | 30 | 37
  Week 9: Monocytes/Leukocytes | -0.16 (2.04) | 0.05 (1.86)
  Week 9: Neutrophils/Leukocytes: number analyzed (Participants) | 30 | 37
  Week 9: Neutrophils/Leukocytes | 0.49 (12.29) | 2.08 (8.89)

8. Secondary Outcome: Mean Change From Baseline in Hemoglobin Levels
Time Frame: Week 9 (end of taper/withdrawal)
Population: Hemoglobin levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 31 | 38
g/dL | -0.06 (0.55) | 0.08 (0.65)

9. Secondary Outcome: Mean Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin Levels
Time Frame: Week 9 (end of taper/withdrawal)
Population: Erythrocyte mean corpuscular hemoglobin levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 31 | 38
pg/cell | 0.13 (0.67) | -0.03 (0.72)

10. Secondary Outcome: Mean Change From Baseline in Erythrocyte Mean Corpuscular Volume Levels
Time Frame: Week 9 (end of taper/withdrawal)
Population: Erythrocyte mean corpuscular volume levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 31 | 38
fL | 0.52 (2.32) | 0.03 (2.39)

11. Secondary Outcome: Number of Patients With Clinically Significant Vital Sign Values
Time Frame: Post-baseline up to 12 weeks
Population: Vital signs were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 45 | 52
Participants
  Increase in weight from baseline >7%: number analyzed (Participants) | 41 | 49
  Increase in weight from baseline >7% | 7 | 13
  Decrease in weight from baseline >7%: number analyzed (Participants) | 41 | 49
  Decrease in weight from baseline >7% | 2 | 2
  Body temperature <36 degrees Celsius | 4 | 6
  Body temperature >38 degrees Celsius | 1 | 0
  Pulse rate <60 beats/min | 1 | 3
  Pulse rate >100 beats/min | 7 | 4
  Respiratory rate <12 breaths/min: number analyzed (Participants) | 43 | 52
  Respiratory rate <12 breaths/min | 0 | 0
  Respiratory rate >20 breaths/min: number analyzed (Participants) | 43 | 52
  Respiratory rate >20 breaths/min | 13 | 17
  Systolic blood pressure <90 mmhg | 5 | 3
  Systolic blood pressure >160 mmhg | 0 | 0
  Diastolic blood pressure <50 mmhg | 3 | 2
  Diastolic blood pressure >120 mmhg | 0 | 0

12. Secondary Outcome: Number of Patients With Clinically Significant Physical Examination Procedure Findings
Description: Number of patients with abnormal physical exam findings are reported.
Time Frame: Baseline up to Day 85 post-baseline
Population: Abnormal physical exam findings were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 49 | 54
Participants
  Abdomen | 2 | 0
  Cardiovascular | 0 | 0
  Chest/lungs | 0 | 0
  Dermatological | 3 | 3
  Endocrine system | 0 | 0
  Gastrointestinal | 0 | 0
  General appearance | 0 | 2
  HEENT | 0 | 1
  Lymphatic | 0 | 0
  Musculoskeletal/Extremities | 0 | 1
  Neurological | 2 | 0
  Other | 0 | 0
  Genitourinary/Reproductive | 0 | 0

13. Secondary Outcome: Number of Patients With Clinically Significant 12-lead Electrocardiogram Findings
Time Frame: Baseline up to Day 85 post-baseline
Population: Clinically significant 12-lead electrocardiogram were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 49 | 54
Participants
  QTcB >450 msec | 7 | 4
  QTcB >480 msec | 2 | 0
  QTcB >500 msec | 1 | 0

14. Secondary Outcome: Number of Participants Reporting Suicidal Ideation or Behavior Using the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS rating scale results since last visit is reported. The presence/absence of any suicidal ideation or behavior is scored based on yes/no responses. The overall number of participants reporting suicidal ideation or behavior is being reported.
Time Frame: Baseline up to Day 92
Population: Suicidal ideation or behavior was assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 49 | 54
Participants
  Suicidal ideation | 4 | 3
  Wish to be dead | 3 | 3
  Non-specific active suicidal thoughts | 2 | 1
  Active suicidal ideation, no intent to act | 1 | 0
  Active suicidal ideation, some intent to act | 0 | 0
  Active suicidal ideation, specific plan/intent | 0 | 0
  Suicidal behavior | 3 | 6
  Actual attempt | 0 | 1
  Interrupted attempt | 0 | 1
  Aborted attempt | 0 | 0
  Preparatory acts or behavior | 0 | 1
  Suicidal behavior item | 0 | 1
  Self-injurious behavior without suicidal intent | 3 | 5
  Completed suicide | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 14 days after last dose, up to approximately 12 weeks.
Arm/Group | GWP42003-P | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/49 | 1/54
Other Adverse Events (participants affected / at risk) | 14/49 | 20/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=49) | Placebo (N=54)
Suicidal ideation (Psychiatric disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=49) | Placebo (N=54)
Headache (Nervous system disorders) | 3 | 4
Pyrexia (General disorders) | 0 | 5
Fatigue (General disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Irritability (Psychiatric disorders) | 0 | 5
Nasopharyngitis (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04745026/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT04745026/SAP_001.pdf